CLINICAL TRIAL: NCT02160262
Title: A Phase 3, 12-Month, Multicenter, Open-label, Flexibly-dosed, Safety Study of SEP 225289 in Adults With Attention Deficit Hyperactivity Disorder (ADHD)
Brief Title: Open-label Safety Study in Adults With ADHD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SEP360-304
Record Dates: First submitted 2014-06-08; First posted 2014-06-10 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-05

CONDITIONS: Adult Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — 4-(3,4-dichlorophenyl)-1,2,3,4-tetrahydronaphthalen-1-amine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dasotraline (Experimental): Dasotraline 4 mg, 6 mg, 8 mg, flexibly dosed
  Interventions: Drug: Dasotraline

INTERVENTIONS:
Drug: Dasotraline — Dasotraline 4 mg, 6 mg, 8 mg, flexibly dosed, once daily

SUMMARY:
To evaluate the long-term safety and tolerability of SEP 225289 in adult subjects with Attention Deficit Hyperactivity Disorder (ADHD)

DETAILED DESCRIPTION:
To evaluate the long-term safety and tolerability of SEP 225289 in adult subjects with ADHD by the incidence of adverse events (AEs; or serious AEs), AEs (or SAEs) leading to discontinuation

ELIGIBILITY:
Inclusion Criteria:

* Subject meets DSM 5 criteria for a primary diagnosis of ADHD (inattentive, hyperactive, or combined presentation) established by a comprehensive psychiatric evaluation that reviews DSM 5 criteria. Diagnosis is confirmed by CAADID Part 2 with checklist for DSM 5.
* Subject has an ADHD RS IV with adult prompts score of ≥ 22 at screening and baseline.
* Subject has agreed to participate by providing written informed consent and is willing and able to comply with the protocol, in the opinion of the investigator.
* Subject is 18 to 55 years old, inclusive, at the time of informed consent.
* Subject is male or a non-pregnant, non lactating female.
* Female subjects must have a negative serum pregnancy test; females who are post menopausal (defined as at least 12 months of spontaneous amenorrhea) and those who have undergone hysterectomy or bilateral oophorectomy will be exempted from the pregnancy test.
* Female subjects of childbearing potential and male subjects with female partners of childbearing potential must agree to use an effective and medically acceptable form of birth control throughout the study period.
* Subject has a negative breath alcohol test and a negative urine drug screen (UDS) for any illicit drug at screening.
* Subject is judged by the investigator to be suitable for participation in a 12 month clinical trial involving open-label dasotraline treatment.
* Subject can read well enough to understand the informed consent form and other subject materials.

Exclusion Criteria:

* Subject has a psychiatric disorder other than ADHD that has been the primary focus of treatment at any time during the 12 months prior to screening.
* Subject has a past history of, or current presentation consistent with, bipolar disorder (including bipolar I and bipolar II), schizophrenia, schizoaffective disorder, or any other psychotic disorder, or a personality disorder per DSM 5 criteria.
* Subject has a history of substance abuse or drug dependence (excluding nicotine and caffeine) within the 12 months prior to screening, as defined by the DSM 5 criteria.
* Subject has a history of epilepsy, seizures (except childhood febrile seizures), unexplained syncope or other unexplained blackouts (except single incident), or head trauma with loss of consciousness lasting more than 5 minutes.
* Subject has a currently active medical condition (other than ADHD) that, in the opinion of the investigator, could interfere with the ability of the subject to participate in the study.
* Subject is currently taking or has taken within the previous 6 months an anticonvulsant medication (eg, phenytoin, carbamazepine, lamotrigine, valproic acid, etc); antipsychotic medication; or lithium (any lithium preparation or formulation).
* Subject is currently taking an alpha 2 adrenergic receptor agonist (including clonidine and guanfacine), or serotonin-norepinephrine reuptake inhibitor (SNRI; eg, venlafaxine), or dopamine-norepinephrine reuptake inhibitor (DNRI; eg, bupropion), or monoamine oxidase [MAO] inhibitor. Note: Subjects who discontinue these medications and wash-out from them for a minimum of 7 days prior to the first dose of study drug will be allowed to enroll in the study.
* Subject is currently undergoing Cognitive Behavioral Therapy (CBT).
* Subject has a Body Mass Index (BMI) less than 18 or greater than 35 kg/m2 (see Appendix V).
* Subject answers "yes" to "Suicidal Ideation" item 4 (active suicidal ideation with some intent to act, without specific plan) or item 5 (active suicidal ideation with specific plan and intent) on the C SSRS assessment at screening (in the past month). Subjects who answer "yes" to this question must be referred to the investigator for follow up evaluation.
* Subject has attempted suicide within 1 year prior to the screening period.
* Subject has history of positive test for Hepatitis B surface antigen or Hepatitis C antibody and has liver function test results at screening above the upper limit of normal for the reference lab.
* Subject is known to have tested positive for human immunodeficiency virus (HIV).
* Subject has a clinically significant abnormality on screening evaluation including physical examination, vital signs, ECG, or laboratory tests that the investigator considers to be inappropriate to allow participation in the study.
* The subject's screening ECG shows a corrected QT interval using Fridericia's formula (QTcF) of ≥ 450 msec for male subjects or ≥ 470 msec for female subjects. Eligibility will be based on the core laboratory ECG interpretation report.
* The subject's screening serum chemistry results show an alanine aminotransferase (ALT) or aspartate aminotransferase (AST) value ≥ 2 times the upper limit of normal (ULN), or a blood urea nitrogen (BUN) value ≥ 1.5 times the ULN for the reference laboratory.
* Subject is currently participating or has participated in a clinical trial within the last 90 days or has participated in more than 2 clinical trials within the past year. This includes studies using marketed compounds or devices.
* Subject has a history of allergic reaction or has a known or suspected sensitivity to any substance that is contained in the study drug formulation.
* Subject has previously been randomized in a clinical trial of dasotraline.
* Subject is likely to be noncompliant in the investigator's opinion.
* Subject is an investigational site staff member or the relative of an investigational site staff member.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 724 (Actual)
Dates: Start 2014-06; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
The incidence of AEs (or SAEs), and AEs (or SAEs) leading to discontinuation. | 12 months

SECONDARY OUTCOMES:
Clinical evaluations (vital signs, physical examination, body weight, and 12 lead ECG) | 12 Months
Clinical laboratory evaluations (serum chemistry, hematology, lipid panel, thyroid panel, and urinalysis) | 12 months
Drug Effects Questionnaire (DEQ) | 12 months
Frequency and severity of suicidal ideation and suicidal behavior using the Columbia - Suicide Severity Rating Scale (C SSRS) | 12 months
Change from baseline in ADHD RS IV with adult prompts total score | 12 months
Change from baseline in Clinical Global Impression - Severity (CGI S) score | 12 months
Change from baseline in the ADHD RS IV with adult prompts inattentiveness and hyperactivity-impulsivity subscale scores | 12 months
Change from baseline in AIM A in global domain scores (Performance and Daily Functioning, Impact of Symptoms: Daily Interference, Impact of Symptoms: Bother/Concern, Relationships/Communication, Living with ADHD, and General Well-being) | 12 months
Change from baseline in Sheehan Disability Scale (SDS) total score | 12 months
Change from baseline in Sheehan Disability Scale (SDS) domain scores: work/school, family life, social life | 12 months
Change from baseline in Behavior Rating Inventory of Executive Function®-Adult Version (BRIEF®) A Global Executive Composite raw score and Behavioral Regulation Index (BRI) raw score and Metacognition Index (MI) raw score. | 12 months
Change from baseline in Pittsburgh Sleep Quality Index (PSQI) global score and 7 component scores. | 12 months
Change from baseline in BRIEF-A Global Executive Composite T-score and BRI T-score and MI T-score. | 12 months
Symptoms of withdrawal using Physician Withdrawal Checklist (PWC) scores, Study Medication Withdrawal Questionnaire (SMWQ) scores, Montgomery-Asberg Depression Rating Scale (MADRS) scores, Hamilton Anxiety Rating Scale (HAM-A) scores | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: SEP289 Medical Director, Study Director — Sumitomo Pharma America, Inc.
Locations (65):
- United States (65):
  - Southern California Research LLC, Beverly Hills, California
  - Pharmacology Research Institute, Encino, California
  - Synergy Clinical Research of Escondido, Escondido, California
  - Collaborative Neuroscience Network, LLC, Garden Grove, California
  - Pharmacology Research Institute, Los Alamitos, California
  - Excell Research, Inc, Oceanside, California
  - Artemis Institute for Clinical Research, San Diego, California
  - MCB Clinical Research Centers, LLC, Colorado Springs, Colorado
  - Florida Clinical Research Center LLC, Bradenton, Florida
  - Gulfcoast Clinical Research, Fort Myers, Florida
  - Broward Research Group, Inc., Hollywood, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Geroge M. Joseph MD, PA, Jacksonville Beach, Florida
  - Compass Research North, LLC, Leesburg, Florida
  - Florida Clinical Research Center, LLC, Maitland, Florida
  - Acumentality, Melbourne, Florida
  - Clinical Neuroscience Solutions, Inc, Orlando, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - Institute for Advanced Medical Research, Alpharetta, Georgia
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - iResearch Atlanta, LLC, Decatur, Georgia
  - Carman Research, Smyrna, Georgia
  - Goldpoint Clinical Research, Indianapolis, Indiana
  - Alpine Clinic, Lafayette, Indiana
  - Psychiatric Associates, Overland Park, Kansas
  - Lake Charles Clinical Trials LLC, Lake Charles, Louisiana
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Rochester Center for Behavioral Medicine, Rochester Hills, Michigan
  - Psychiatric Care & Research Center, O'Fallon, Missouri
  - Midwest Research Group, Saint Charles, Missouri
  - Premeir Psychiatric Research Institute, LLC, Lincoln, Nebraska
  - Center for Psychiatry and Behavioral Medicine, Inc., Las Vegas, Nevada
  - Center for Emotional Fitness, Cherry Hill, New Jersey
  - Bioscience Research, Mount Kisco, New York
  - Village Clinical Research Inc., New York, New York
  - NYU School of Medicine, New York, New York
  - Medical & Behavioral Health Research, New York, New York
  - The Medical Research Network, LLC, New York, New York
  - Fieve Clinical Research, New York, New York
  - Woodhull Medical & Mental Health Center, Staten Island, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - Duke University Medical Center, Durham, North Carolina
  - Neuro-Behavioral Clinical Research, Canton, Ohio
  - Midwest Clinical Research Center, Dayton, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Cutting Edge Research Group, Oklahoma City, Oklahoma
  - Summit Research Network, Portland, Oregon
  - Oregon Center for Clinical Investigations, Inc., Portland, Oregon
  - Suburban Research Associates, Media, Pennsylvania
  - Keystone Clinical Studies, LLC, Norristown, Pennsylvania
  - Sleep Diagnosists and Treatment Centers, West Chester, Pennsylvania
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Clinical Neuroscience Solutions, Memphis, Tennessee
  - Research Strategies of Memphis, LLC, Memphis, Tennessee
  - FutureSearch Trials of Dallas, LP, Dallas, Texas
  - Pillar Clinical Research, LLC, Dallas, Texas
  - Houston Clinical Trials, LLC, Houston, Texas
  - Clinical Trials of Texas, Inc, San Antonio, Texas
  - Family Psychiatry of the Woodlands, The Woodlands, Texas
  - Neuropsychiatric Associates, Woodstock, Vermont
  - NeuroScience, Inc, Herndon, Virginia
  - Summit Research Network (Seattle) LLC, Seattle, Washington
  - Dean Foundation, Middleton, Wisconsin
  - Eastside Therapeutic Resource, Middleton, Wisconsin